CLINICAL TRIAL: NCT00212095
Title: Phase II Study of Docetaxel Combined With Ketoconazole in the First-line Treatment of Locally Advanced or Metastatic Breast Cancer Patients With Measurable Primary Breast Tumor
Brief Title: Docetaxel Combined With Ketoconazole in Treatment of Breast Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National University Hospital, Singapore (Other)
Responsible Party: Principal Investigator, Haematology-Oncology, Senior Consultant, National University Hospital, Singapore
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BR01/07/05
Record Dates: First submitted 2005-09-13; First posted 2005-09-21 (Estimated); Last update posted 2012-11-01 (Estimated); Status verified 2012-10

CONDITIONS: Metastatic Breast Cancer
Keywords: breast cancer; docetaxel; gene expression; proteomics
MeSH Terms: conditions — Breast Neoplasms | interventions — Docetaxel; Ketoconazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- docetaxel and ketoconazole (Experimental)
  Interventions: Drug: docetaxel and ketoconazole

INTERVENTIONS:
Drug: docetaxel and ketoconazole — Docetaxel will be obtained locally from the manufacturer. Storage conditions for unopened vials, reconstitution, and storage conditions for the reconstituted solution will follow the manufacturer's recommendations. Docetaxel solutions should be prepared and stored in glass, polypropylene or polyolefin containers. Non-PVC containing and polyethylene-lined administration sets should be used.
  Ketoconazole is available commercially in 200 mg tablet. Ketoconazole is to be administered at a dose of 200mg BID orally for six doses, starting two days before docetaxel administration. The fifth dose should be administered on the day of and before administering docetaxel, while the sixth dose should be administered in the evening of the day of docetaxel administration.

SUMMARY:
Patients with locally advanced or metastatic breast cancer and with measurable primary breast tumor will be treated with 70mg docetaxel combined with ketoconazole. Serial tumor biopsies and plasma samples will be taken for gene expression and proteomics studies to identify biomarkers that may predict for treatment response.

DETAILED DESCRIPTION:
We hypothesize that 70mg docetaxel co-administered with ketoconazole would result in similar clinical efficacy as conventional doses of docetaxel (75mg/m2 body surface area) in terms of clinical and pathological response rates in metastatic breast cancer. We further hypothesize that tumor genomic and proteomic changes and serum proteomic changes would correlate with tumor response. We are also looking to correlate drug pharmacokinetics with treatment toxicity, genotype of drug metabolizing enzymes and transporters, and peripheral mononuclear cell gene expression profiles. The primary objectives are to evaluate the clinical response rate of 70mg docetaxel with ketoconazole in metastatic breast cancer, and to evaluate the pathological response rate in the primary tumor following four cycles of docetaxel and ketoconazole.

ELIGIBILITY:
Inclusion Criteria:

* Female, age >= 18 years.
* Histologic or cytologic diagnosis of breast carcinoma.
* T3-4 breast cancer with measurable primary breast tumor, defined as palpable tumor with both diameters 2.0cm or greater as measured by caliper.
* Patients must not have received prior chemotherapy or hormonal therapy for the treatment of breast cancer.
* Karnofsky performance status of 70 or higher.
* Estimated life expectancy of at least 12 weeks.
* Adequate organ function including the following:

  - Bone marrow: Absolute neutrophil (segmented and bands) count (ANC) >= 1.5 x 109/L Platelets >= 100 x 109/L

  - Hepatic: Bilirubin <= 1.5 x upper limit of normal (ULN), ALT or AST <= 2.5x ULN, (or <5 X with liver metastases)

  - Renal: creatinine <= 1.5x ULN
* Left ventricular ejection fraction >=50%
* Signed informed consent from patient or legal representative.
* Patients with reproductive potential must use an approved contraceptive method if appropriate (eg, intrauterine device, birth control pills, or barrier device) during and for three months after the study. Females with childbearing potential must have a negative serum pregnancy test within 7 days prior to study enrollment.

Exclusion Criteria:

* Prior treatment for locally advanced or metastatic breast cancer.
* Treatment within the last 30 days with any investigational drug.
* Concurrent administration of any other tumor therapy, including cytotoxic chemotherapy, hormonal therapy, and immunotherapy.
* Active infection that in the opinion of the investigator would compromise the patient's ability to tolerate therapy.
* Pregnancy.
* Breast feeding.
* Serious concomitant disorders that would compromise the safety of the patient or compromise the patient's ability to complete the study, at the discretion of the investigator.
* Poorly controlled diabetes mellitus.
* Second primary malignancy that is clinically detectable at the time of consideration for study enrollment.
* Symptomatic brain metastasis.
* History of significant neurological or mental disorder, including seizures or dementia.
* Peripheral neuropathy of CTC grade 2 or above (NCI CTC version 3).
* History of hypersensitivity to drugs formulated in Tween 80, the vehicle used for commercial docetaxel formulations.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2005-06; Primary Completion 2007-04 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
1. Evaluate the clinical response rate of 70mg docetaxel with ketoconazole in metastatic breast cancer. | 4 months
2. Evaluate the pathological response rate in the primary tumor following four cycles of docetaxel and ketoconazole. | 5 months

SECONDARY OUTCOMES:
1. To study tumor genomics and proteomics and serum proteomics in breast cancer in response to docetaxel/ketoconazole. | 2 years
2. To compare tumor genomics and proteomics and serum proteomics in breast cancer in response to docetaxel/ketoconazole to that induced by docetaxel alone in a prior study (HO B17/02). | 2 years
3. To correlate docetaxel pharmacokinetics with (1)Genetic polymorphisms of drug metabolizing enzymes(2)Drug toxicity & tumor response(3)Peripheral mononuclear cell gene expression profiles | 3 years
(4) To study ondansetron pharmacokinetics and correlate that with genetic polymorphisms | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Soo-Chin Lee, MD, Principal Investigator — Consultant
Locations (1):
- National University Hospital, Singapore, Singapore

REFERENCES:
- [Derived] Lim YW, Goh BC, Wang LZ, Tan SH, Chuah BYS, Lim SE, Iau P, Buhari SA, Chan CW, Sukri NB, Cordero MT, Soo R, Lee SC. Pharmacokinetics and pharmacodynamics of docetaxel with or without ketoconazole modulation in chemonaive breast cancer patients. Ann Oncol. 2010 Nov;21(11):2175-2182. doi: 10.1093/annonc/mdq230. Epub 2010 Apr 29. PMID 20430905